CLINICAL TRIAL: NCT01849341
Title: Clinical Trial Phase III Blind, Parallel Group to Analyze Differences in the Safety of Roflumilast Administered Once a Day on Alternate Days for Two Weeks Compared to the Usual Dosage Once Daily
Brief Title: Roflumilast Safety Administered Once a Day on Alternate Days for Two Weeks Compared to the Usual Dosage Once Daily
Acronym: ROFLU2011
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: ROFLU2011
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Roflumilast alternated days (Experimental): Intervention: 500 mcg per day on alternate days (roflumilast 500μg eod) for 2 weeks
  Interventions: Drug: Roflumilast alternated days
- Roflumilast 500 mcg per day (Active Comparator): Roflumilast 500μg standard dosage
  Interventions: Drug: Roflumilast 500 mcg per day

INTERVENTIONS:
Drug: Roflumilast alternated days — 500 mcg per day on alternate days (roflumilast 500μg eod) for 2 weeks
  Other Names: schedule change
  Arms: Roflumilast alternated days
Drug: Roflumilast 500 mcg per day
  Other Names: Standard dosage
  Arms: Roflumilast 500 mcg per day

SUMMARY:
It is a phase IV clinical trial: longitudinal, prospective, evaluator-blind, randomized into 2 groups of patients with chronic obstructive pulmonary disease (COPD). The intervention group was based on the administration of roflumilast 500 mcg per day on alternate days (roflumilast 500μg eod) for 2 weeks (phasing). In the control group assigned to undertake the treatment according to the standard dosage (roflumilast 500μg od).

The patient monitoring will be done by one of the sub-investigators fully independent team that started the medication keeping the pattern masking by single blind, and since it aims to assess the frequency of adverse events (AEs) in both groups were collected systematically different AEs and their characteristics at 15 days (V1), and from that moment a month (V2) and 2 months (V3). Likewise, other data collected (functional demographic, comorbidities, home treatment, anxiety and depression and quality of life).

The purpose of this study is to assess whether the administration of roflumilast by a gradual pattern varies the incidence of discontinuations due to adverse events when compared with the usual dosage.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD in severe degree GOLD criteria, assessed by post-bronchodilator spirometry (FEV1 <50%, FEV1/Forced vital capacity (FVC) <70% of theory).
* Age over 18 years.
* Productive cough recurrently most days for at least three months a year and at least 2 consecutive years.
* History from smoking prior> 15 to 20 packs / year.
* An exacerbation in the previous year.
* Stability clinic in the last 30 days.

Exclusion Criteria:

* Pregnancy / breastfeeding.
* Acute infections.
* Patients with severe mental disorder or uncontrolled, in the opinion of the investigator, would make the patient has a higher risk due to their participation in the study, could be a confounding factor in the study's results or is likely to prevent that the patient meets the requirements of the study or to complete the study.
* Patients cachectic or the risk of cachexia.
* HIV infection.
* Severe immune Infections (systemic lupus erythematosus, multiple sclerosis, etc.).
* Gastroesophageal reflux symptoms and diagnosis established.
* Hiatal hernia.
* Peptic ulcer disease.
* Inflammatory bowel pathology.
* Neoplastic pathology: current diagnosis of cancer other than basal cell or squamous cell carcinoma of the skin.
* Moderate to severe hepatic impairment (Child-Pugh BC).
* Inability to understand / perform the techniques.
* Home treatment with theophylline, methotrexate, azathioprine, infliximab, etanercept, inducers of cytochrome P450 (eg, rifampicin, phenobarbital, carbamazepine, phenytoin),cytochrome P450 3A4 (CYP3A4) inhibitors (erythromycin and ketoconazole), oral contraceptives (gestodene and ethinyl estradiol), making prolonged oral corticosteroids, or a drug that contains fluvoxamine, enoxacin and cimetidine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Difference of Adverse Events | 2 weeks
  Difference in the proportion of patients who leave the study for AEs between the control group (roflumilast 500μg od) and intervention (roflumilast 500μg eod)

SECONDARY OUTCOMES:
Patients who leave the study | two weeks
  Difference in the proportion of patients who leave the study for AEs between the control group (roflumilast 500μg od) alternating pattern (in patients with impaired tolerance) and intervention (roflumilast 500μg eod) between visits V2 and V0.

CONTACTS AND LOCATIONS:
Overall Officials: Teodoro Montemayor Rubio, M.D. Ph D, Study Chair — Hospital Universitario Virgen Macarena; Ruth Ayerbe, M.D, Principal Investigator — Complejo Hospitalario de Especialidades Juan Ramón Jimenez; Gregorio Soto, M.D., Principal Investigator — Hospital de Jerez; Francisco L Muñoz, M.D., Principal Investigator — Hospital Universitario Reina Sofía; Concepción Morales, M.D., Principal Investigator — H.U. Virgen de las Nieves; José L de la Cruz, M.D., Principal Investigator — Complejo Hospitalario Carlos Haya; Cristina García, M.D., Principal Investigator — Hospital Universitario de Puerto Real; Bernardino Alcázar, M.D., Principal Investigator — HAR de Loja; Rosa Vazquez, M.D., Principal Investigator — Hospital Infanta Elena
Locations (4):
- Spain (4):
  - Hospital de Jerez, Jerez de la Frontera, Cádiz
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - H.U. Virgen de las Nieves, Granada, Granada
  - Hospital Universitario Virgen Macarena, Seville, Sevilla